CLINICAL TRIAL: NCT02200835
Title: Gender-related Differences in Chinese Patients With AAD
Status: Completed | Type: Observational
Sponsor: General Hospital of Beijing PLA Military Region (Other)
Responsible Party: Principal Investigator, Yang Li, Dr., General Hospital of Beijing PLA Military Region
Other Study IDs: GHBeijing-20140701; GDAAD-20140701
Record Dates: First submitted 2014-07-24; First posted 2014-07-25 (Estimated); Last update posted 2014-07-25 (Estimated); Status verified 2014-01

CONDITIONS: Aneurysm Dissecting
Keywords: aortic dissection; Chinese patients; gender differences
MeSH Terms: conditions — Aortic Dissection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Few data exist on gender-related differences in clinical features, management, and outcomes of acute aortic dissection (AAD) in China. Accordingly, we enrolled 2015 patients with AAD from 15 hospitals in China to access differences in clinical features, management and outcomes between men and women. in this study, our results provided new insights into gender-related differences in clinical features, management and outcomes in the Chinese patients with AAD. Important implications may be helpful to improve diagnostic and therapeutic outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute aortic dissection

Exclusion Criteria:

* Simple dilated aneurysm and penetrating atherosclerotic ulcer

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Chinese pupolation and foreign citizen of Chinese origin from 15 major hospitals in China
Sampling Method: Probability Sample
Enrollment: 2015 (Actual)
Dates: Start 2012-01; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
all patients with acute aortic dissection | 2 years